CLINICAL TRIAL: NCT07382102
Title: The Impact of Nutrition Education on Nursing Students' Nutrition Knowledge, Attitudes, Physical Activity, and Sleep Quality
Brief Title: Effect of Nutrition Education on Nursing Students' Health Behaviors and Sleep Quality
Acronym: NUTRI-SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AICU-NUTRITION-01
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Health-related Behaviors in Nursing Students; Nutrition and Sleep Behaviors
Keywords: Nutrition education; Dietary behavior; Nursing students; Physical activity; Sleep quality
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: All participants receive the same nutrition education intervention and are evaluated before the intervention, immediately after completion, and three months after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Education Intervention (Experimental): Participants in this single-arm study received a structured nutrition education program designed to improve nutrition knowledge, dietary behaviors, physical activity awareness, and sleep-related lifestyle habits. The education program was delivered over multiple sessions and covered basic nutrition principles, food groups, balanced diet concepts, healthy food choices, and the relationship between nutrition, physical activity, and sleep. All participants received the same intervention.
  Interventions: Behavioral: Nutrition Education Program

INTERVENTIONS:
Behavioral: Nutrition Education Program — A structured nutrition education program delivered through multiple educational sessions. The intervention focuses on improving nutrition knowledge, healthy food choices, balanced diet principles, and awareness of the relationship between nutrition, physical activity, and sleep. The program is educational in nature and does not involve medications, medical devices, or invasive procedures.

SUMMARY:
This study aims to evaluate the effects of a structured nutrition education program on nursing students' nutrition knowledge, dietary behaviors, physical activity levels, and sleep quality. University students, particularly those studying in health-related fields, often experience irregular eating habits, insufficient physical activity, and poor sleep quality due to academic workload and lifestyle factors. These behaviors may negatively affect both their personal health and their future professional roles.

In this study, nursing students will participate in a multi-session nutrition education program designed to improve awareness of healthy eating, balanced diets, and lifestyle behaviors. Data will be collected before the education program, immediately after completion, and three months later. Outcomes will include changes in nutrition knowledge, food choices, physical activity levels, and sleep quality.

The results of this study are expected to contribute to the development of effective educational strategies that promote healthy lifestyle behaviors among nursing students and support their well-being during university education.

DETAILED DESCRIPTION:
This interventional study is designed to examine the impact of a structured nutrition education program on nursing students' health-related behaviors, including nutrition knowledge, dietary attitudes and behaviors, physical activity level, and sleep quality. Nursing students represent a critical population, as they are future health professionals who will play an important role in health promotion and patient education. However, during university education, nursing students may develop unhealthy eating patterns, low physical activity levels, and poor sleep quality due to academic demands and lifestyle changes.

The study will be conducted at the Faculty of Health Sciences, Department of Nursing, at Ağrı İbrahim Çeçen University. Eligible participants include undergraduate nursing students who have not previously received formal nutrition education and who voluntarily agree to participate in the study.

The intervention consists of a structured nutrition education program delivered over multiple sessions. The education content includes basic nutrition principles, food groups, balanced diet concepts, healthy food choices, nutrition-health relationships, and lifestyle factors related to physical activity and sleep. The education program is designed to increase awareness and encourage healthier behaviors rather than to provide clinical treatment.

Data collection will occur at three time points: before the intervention (baseline), immediately after completion of the nutrition education program, and three months after the intervention to assess the sustainability of potential changes. Data collection tools include questionnaires assessing sociodemographic characteristics, nutrition knowledge, dietary behaviors, food consumption frequency, physical activity level, and sleep quality. Physical activity will be evaluated using a standardized physical activity questionnaire, and sleep quality will be assessed using a validated sleep quality index.

The primary objective of the study is to assess changes in nutrition knowledge following the education program. Secondary objectives include evaluating changes in dietary behaviors, physical activity level, and sleep quality over time. Statistical analyses will be conducted to compare outcomes across the three measurement points.

This study involves minimal risk to participants. The intervention is educational in nature and does not include invasive procedures, medications, or medical devices. Ethical approval has been obtained from the institutional ethics committee, and informed consent will be obtained from all participants prior to data collection. The findings of this study are expected to provide evidence supporting the integration of structured nutrition education into nursing curricula to promote healthy lifestyle behaviors among students.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students enrolled at the Faculty of Health Sciences.
* Aged between 18 and 30 years.
* Have not previously received formal nutrition education.
* Able to read and understand the study questionnaires.
* Willing to participate and provide informed consent.

Exclusion Criteria:

* Having previously received structured or formal nutrition education.
* Presence of a medical condition that affects dietary intake or sleep patterns.
* Use of medications that significantly influence appetite, metabolism, or sleep.
* Unwillingness or inability to complete the study questionnaires.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition Knowledge Score | Baseline, immediately after completion of the nutrition education program, and 3 months after the intervention
  Nutrition knowledge is measured using a structured Nutrition Knowledge Questionnaire developed for nursing students. The questionnaire produces a total score ranging from 0 to 100 points, with higher scores indicating higher nutrition knowledge. Changes in total nutrition knowledge scores across the three time points are analyzed.

SECONDARY OUTCOMES:
Change in Dietary Behavior Scores | Baseline; immediately after completion of the nutrition education program; 3 months after the intervention
  Dietary behaviors are assessed using Food Choice and Dietary Behavior Questionnaires, including food frequency assessment.
  The questionnaires yield a total dietary behavior score ranging from 0 to 100, with higher scores indicating healthier dietary behaviors.
  Frequency-based measures are reported as times per day/week.
Change in Physical Activity Level | Baseline, immediately after completion of the nutrition education program, and 3 months after the intervention
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI). The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. Changes in total and subscale scores over time are analyzed.
Change in Sleep Quality Score | Baseline, immediately after completion of the nutrition education program, and 3 months after the intervention
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI). The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. Changes in total and subscale scores over time are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Faculty of Health Sciences Department of Nursing, Ağrı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small sample of nursing students and includes potentially identifiable educational and lifestyle information. Data were collected solely for the purposes of this study, and participant confidentiality and privacy cannot be fully ensured with data sharing. Aggregate data only will be reported in publications.

REFERENCES:
- [Background] Hamulka J, Wadolowska L, Hoffmann M, Kowalkowska J, Gutkowska K. Effect of an Education Program on Nutrition Knowledge, Attitudes toward Nutrition, Diet Quality, Lifestyle, and Body Composition in Polish Teenagers. The ABC of Healthy Eating Project: Design, Protocol, and Methodology. Nutrients. 2018 Oct 5;10(10):1439. doi: 10.3390/nu10101439. PMID 30720795
- [Background] Mangwane QEM, Egal A, Oosthuizen D. Impact of a Nutrition Knowledge Intervention on Knowledge and Food Behaviour of Women Within a Rural Community. Nutrients. 2024 Nov 28;16(23):4107. doi: 10.3390/nu16234107. PMID 39683501
- [Background] Bajamal E, Alotaibi J, Balamash D, Alsaeedi E, Ali H, Alzahrani J, Swat L, Alamri A, Jundi R, Alzahrani R, Alharbi S. The Association Between Physical Activity and Quality of Sleep Among Nursing Students in Saudi Arabia. Healthcare (Basel). 2025 Aug 14;13(16):1991. doi: 10.3390/healthcare13161991. PMID 40868607
- [Background] Zaghamir DEF, Ibrahim AM. Efficiency of an intervention study on nursing students' knowledge and practices regarding nutrition and dietary habits. Libyan J Med. 2023 Dec;18(1):2281121. doi: 10.1080/19932820.2023.2281121. Epub 2023 Nov 17. PMID 37976204